CLINICAL TRIAL: NCT03850509
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Proof-of-Concept Trial to Assess the Efficacy and Safety of Orally Administered OPS-2071 for 12 Weeks in Subjects With Crohn's Disease Showing Symptoms of Active Inflammation Despite Ongoing Treatment
Brief Title: Efficacy and Safety of Oral OPS-2071 in Participants With Crohn's Disease Showing Symptoms of Active Inflammation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 341-201-00004; 2019-000176-41 (EudraCT Number)
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Inflammatory bowel disease; Fluoroquinolones; Inflammation; Intestine; Digestive tract; Abdominal pain; Diarrhea
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Inflammation; Abdominal Pain; Diarrhea

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two or more parties are unaware of the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OPS-2071 150 mg BID (Experimental): Participants were to receive OPS-2071 150 mg, tablets, orally, twice daily (BID) in the morning and evening (8 to 12 hours apart) with 240 milliliters (mL) of water for up to 12 weeks.
  Interventions: Drug: OPS-2071
- OPS-2071 300 mg BID (Experimental): Participants received OPS-2071 300 mg, tablets, orally, BID in the morning and evening (8 to 12 hours apart) with 240 mL of water for up to 6 weeks.
  Interventions: Drug: OPS-2071
- OPS-2071 600 mg BID (Experimental): Participants were to receive OPS-2071 600 mg, tablets, orally, BID in the morning and evening (8 to 12 hours apart) with 240 mL of water for up to 12 weeks.
  Interventions: Drug: OPS-2071
- Placebo (Placebo Comparator): Participants received OPS-2071-matched placebo, tablets, orally, BID in morning and evening (8 to 12 hours apart) with 240 mL of water for up to 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPS-2071 — OPS-2071 300 mg, tablets, orally, BID.
  Arms: OPS-2071 150 mg BID; OPS-2071 300 mg BID; OPS-2071 600 mg BID
Drug: Placebo — OPS-2071-matched placebo, tablets, orally, BID.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects and safety of OPS-2071 (150, 300, or 600 mg twice a day [BID]) versus placebo, as add-on therapy in participants with Crohn's disease who show symptoms of active inflammation despite being on ongoing treatment.

DETAILED DESCRIPTION:
OPS-2071 is a novel agent that is currently being developed for the treatment of Crohn's disease and was previously investigated for the treatment of enteric infection, including those caused by Clostridium difficile. OPS-2071 belongs to the fluoroquinolone family of compounds and has shown anti-inflammatory and potent antibacterial activity in in vitro and in vivo assays. OPS-2071 is anticipated to be effective in the treatment of Crohn's disease due to its unique mode of action. In vitro investigations of OPS-2071 showed a dual mechanism of action, including a potent, broad spectrum antibacterial effect and a strong anti-inflammatory effect that translated into significant attenuation of numerous cytokines, including TNF-alpha (TNF-α) screening.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 and 70 years, inclusive
* Diagnosis of Crohn's disease localized in the ileum and/or colon, with active mucosal inflammation and visible lesion(s), documented by centrally read ileocolonoscopy and a Simple Endoscopic Score for Crohn's Disease (SES-CD) ≥ 6 (≥ 4 for isolated ileal disease).
* Participants who do not have an optimal response (daily stool frequency > 3 and pain score > 1) to their current ongoing treatment of biologics (eg, first anti-tumor necrosis factor-alpha [TNF-α] monoclonal antibody), immunosuppressants, low-dose steroids, or 5-aminosalicylic acid (5-ASA) formulations.
* Participants who are on stable Crohn's disease medications for at least 4 weeks.
* Participants with a CDAI score between 180 and 450 points, inclusive.
* Participants who are willing and able to follow the trial protocol and have signed informed consent.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving IMP.
* Sexually active males or WOCBP who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of IMP. If employing birth control, 2 of the following precautions must be used: vasectomy, tubal ligation, intrauterine device, birth control pill, birth control implant, or birth control depot injection. A vaginal diaphragm, condom with spermicide, or sponge with spermicide may also be used as measures to prevent pregnancy, but must be used in combination with at least one of the previous methods.
* Participants taking any nonsteroidal anti-inflammatory drugs that cannot be stopped or replaced.
* Use of prednisone or prednisolone > 30 mg/day or budesonide > 9 mg/day within 4 weeks prior to screening; or intravenous steroids within 4 weeks prior to screening.
* Participants taking antithrombotic drugs.
* Participants with symptomatic bowel stenosis, fistula, or stoma; or with more than 2 bowel resections.
* Participants with short bowel syndrome.
* participants with known existing aortic aneurysm, or who are at risk for an aortic aneurysm, such as participants with peripheral atherosclerotic vascular diseases, uncontrolled hypertension, certain genetic conditions such as Marfan syndrome and Ehlers-Danlos syndrome, and elderly participants (over the age of 70).
* Participants with known or suspected (family history, unexplained syncope) long QT syndrome or QTcF > 470 msec for females or > 450 msec for males at baseline.
* Participants with inadequate organ function, as follows:

  * Serum creatinine > 1.5x the upper limit of normal (ULN)
  * Aspartate aminotransferase or alanine aminotransferase levels > 1.5x ULN
  * Total bilirubin > 1.5x ULN. Elevated unconjugated bilirubin related to Gilbert's syndrome is allowed.
* Use of antibiotics (eg. metronidazole, rifaximin, tinidazole, ciprofloxacin, clarithromycin) within 15 days prior to screening or for greater than 2 months within the past year. A short course (maximum of 5 days) of antibiotics will be permitted during the trial, as needed, for indications other than Crohn's disease.
* Known hypersensitivity to quinolones or other significant adverse reaction to quinolones.
* Conditions or circumstances that could prevent completion of the trial according to the judgment of the investigator, including an uncontrolled comorbidity, heart condition, or dysfunction of any other organ; peripheral neuropathy; known arrhythmias, atrial fibrillation, or paroxysmal tachycardia; history of myasthenia gravis; history of drug or alcohol abuse, mental illness, or noncompliance with treatments or visits; or known immune-deficiency.
* HIV infection, viral hepatitis, prior organ transplant, or malignant disease that is not in remission for at least 3 years, with the exception of basal cell carcinoma.
* Participants who have used any investigational drug within 2 months prior to screening.
* Blood donation in the last 2 months.
* Use of inhibitors of UGT1A1 and UGT1A9 (eg, Silybin, diclofenac, mycophenolic acid, efavirenz, regorafenib) and BCRP (eg, Estrone, 17β-estradiol, flavonoids, herb extracts, gefitinib, imatinib, tamoxifen, novobiocin, nelfinavir, ritonavir, dipyridamole, fumitremorgin C, Ko143, cyclosporine, curcumin, eltrombopag, omeprazole, ivermectin).
* Participants with a history of treatment failure with 2 or more biologics.
* Participants with risk factors for tendon rupture (ie, psoriasis, ankylosing spondylitis, competitive athletes, renal failure, diabetes mellitus) or who have a history of tendon rupture and/or ongoing tendinopathy.
* Participants with systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg.
* Participants taking quinidine, procainamide, disopyramide, encainide, flecainide, sotalol, amiodarone, ibutilide, dronedarone, or propafenone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (24):
  - United States, California, Los Angeles, California
  - United States, California, San Carlos, California
  - United States, Colorado, Colorado Springs, Colorado
  - United States, Florida, Clearwater, Florida
  - United States, Florida, Hialeah, Florida
  - United States, Florida, Kissimmee, Florida
  - United States, Florida, Naples, Florida
  - United States, Florida, Orlando, Florida
  - United States, Florida, Plantation, Florida
  - United States, Georgia, Decatur, Georgia
  - United States, Georgia, Doraville, Georgia
  - United States, Kansas, Shawnee Mission, Kansas
  - United States, Maryland, Chevy Chase, Maryland
  - United States, North Carolina, Greenville, North Carolina
  - United States, Ohio, Cincinnati, Ohio
  - United States, Ohio, Dayton, Ohio
  - United States, Oklahoma, Oklahoma City, Oklahoma
  - United States, South Carolina, Rock Hill, South Carolina
  - United States, Texas, Austin, Texas
  - United States, Texas, Harlingen, Texas
  - United States, Texas, San Antonio, Texas
  - United States, Texas, Sugar Land, Texas
  - United States, Texas, Tyler, Texas
  - United States, Virginia, Lynchburg, Virginia
- Poland (5):
  - Poland, Knurów
  - Poland, Lodz
  - Poland, Oświęcim
  - Poland, Poznan
  - Poland, Rzeszów

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 2 investigative sites in the United States and Poland from 25 February 2020 to 22 May 2020.
Pre-assignment Details: Participants with Crohn's disease showing symptoms of active inflammation despite ongoing treatment were enrolled and randomized in this study to receive OPS-2071 300 mg BID and OPS-2071 matched placebo. Participants were also to be randomized in OPS-2071 150 mg and 600 mg, however, the study was terminated before the enrollment of participants in the respective arms.
Groups:
- OPS-2071 300 mg BID: Participants received OPS-2071 300 mg, tablets, orally, twice daily (BID) in the morning and evening (8 to 12 hours apart) with 240 milliliters (mL) of water for up to 6 weeks.
Period: Overall Study
Arm/Group | OPS-2071 300 mg BID | Placebo
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study Terminated by the Sponsor (Due to COVID-19 Situation) | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized Set included all participants who were randomized into this trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | OPS-2071 300 mg BID | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Clinical Remission Based on Crohn's Disease Activity Index (CDAI) Score
Description: Clinical remission was defined as CDAI score <150 at Week 12. The CDAI evaluated severity of signs and symptoms of Chron's Disease. Some components of the CDAI were reported by the investigator (physical examination for the presence of an abdominal mass and extraintestinal complications, laboratory results for hematocrit levels, and weight) while other components were determined with data collected in a participant diary (number of liquid or soft stools, number of antidiarrheal medications, abdominal pain score, and general well-being). The index values of 150 and below were associated with quiescent disease; values above that indicated active disease, values >=220 indicated moderate to severe disease, and values above 450 were seen with extremely severe disease.
Time Frame: Week 12
Population: This outcome measure was not analyzed as no participants reached Week 12 time point due to early termination of the study.
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Endoscopic Response Based on Simple Endoscopic Score for Crohn's Disease (SES-CD)
Description: Endoscopic response was defined as a reduction of the SES-CD by at least 50%, at Week 12. The SES-CD is a total score that indicates endoscopic disease activity status based on endoscopy results regarding the size of ulcers, surface ulceration, affected surface size, and presence of luminal narrowing. Each item is scored from 0-3, with total score from 0-60 . Higher score indicates more severe endoscopic activity.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change From Baseline in the SES-CD Score at Week 12
Description: The SES-CD is a total score that indicates endoscopic disease activity status based on endoscopy results regarding the size of ulcers, surface ulceration, affected surface size, and presence of luminal narrowing. Each item is scored from 0-3, with a total score from 0-60. A higher score indicates more severe endoscopic activity. A negative change from baseline indicates improvement.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 1
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Two-item Participant Reported Outcome (PRO-2) Remission
Description: PRO-2 remission was defined as stool frequency =< 3 times per day and abdominal pain =< 1 at Week 12. The PRO-2 is a symptom control measure based on 2 participant-reported components (stool frequency and abdominal pain) of the CDAI (on an 11-point scale where 0=no pain to 10=worst imaginable pain). A weekly score was calculated for the liquid or soft stool frequency and a separate weekly score was calculated for abdominal pain, in each case based on daily symptom reporting. PRO2 is a composite index consisting of weighted scoring of both variables. PRO2 scores ranges from 0 to approximately 45, higher score indicates higher disease activity.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With Clinical Response Based on CDAI Score
Description: Clinical response was defined as at least a 25% decrease in the CDAI score at Week 12. The CDAI evaluated the severity of signs and symptoms of Chron's Disease. Some components of the CDAI were reported by the investigator (physical examination for the presence of an abdominal mass and extraintestinal complications, laboratory results for hematocrit levels, and weight) while other components were determined with data collected in a participant diary (number of liquid or soft stools, number of antidiarrheal medications, abdominal pain score, and general well-being). The index values of 150 and below were associated with quiescent disease; values above that indicated active disease, values >=220 indicated moderate to severe disease, and values above 450 were seen with extremely severe disease.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Endoscopic Remission Based on SES-CD
Description: Endoscopic remission was defined as an SES-CD total score of 0 to 2; or a score of 0 to 4, with no individual subscore greater than 1 at Week 12. The SES-CD is a total score that indicates endoscopic disease activity status based on endoscopy results regarding the size of ulcers, surface ulceration, affected surface size, and presence of luminal narrowing. Each item is scored from 0-3, with a total score from 0-60. A higher score indicates more severe endoscopic activity.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With a Decrease in the CDAI Score at Week 12
Description: Percentage of participants who had a decrease of at least => 100 points in CDAI scores were to be reported. The CDAI evaluated the severity of signs and symptoms of Chron's Disease. Some components of the CDAI were reported by the investigator (physical examination for the presence of an abdominal mass and extraintestinal complications, laboratory results for hematocrit levels, and weight) while other components were determined with data collected in a participant diary (number of liquid or soft stools, number of antidiarrheal medications, abdominal pain score, and general well-being). The index values of 150 and below were associated with quiescent disease; values above that indicated active disease, values >=220 indicated moderate to severe disease, and values above 450 were seen with extremely severe disease.
Time Frame: Week 12
Population: as for outcome 1
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant and that does not necessarily have a causal relationship with the treatment. An SAE is defined as any fatal; life-threatening; persistently or significantly disabling or incapacitating; required in-patient hospitalization or prolonged hospitalization; a congenital anomaly/birth defect; or other medically significant event that, based upon appropriate medical judgment, may have jeopardized the subject and may have required medical or surgical intervention. A TEAE is defined as an AE that occurred after the administration of investigational medicinal product (IMP).
Time Frame: From the signing of the informed consent form up to early termination (up to approximately 9 weeks)
Population: Safety Population included all participants who were administered at least one dose of IMP.
Measure: Number; unit: percentage of participants
Arm/Group | OPS-2071 300 mg BID | Placebo
Number analyzed (Participants) | 2 | 1
percentage of participants | 50.0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form up to early termination (up to approximately 9 weeks)
Description: Safety Analysis Set (SAS) population included all participants who were administered at least one dose of the investigational medicinal product (IMP).
Arm/Group | OPS-2071 300 mg BID | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPS-2071 300 mg BID (N=2) | Placebo (N=1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT03850509/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03850509/SAP_001.pdf